CLINICAL TRIAL: NCT03557567
Title: NGS Strategy Effectiveness in Molecular Diagnosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Regione Emilia-Romagna (Other)
Responsible Party: Sponsor
Other Study IDs: PRUA1GR-2013-00000177
Record Dates: First submitted 2018-05-18; First posted 2018-06-15 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Multiple Osteochondroma; Osteogenesis Imperfecta
MeSH Terms: conditions — Exostoses, Multiple Hereditary; Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MO patients
  Interventions: Diagnostic Test: NGS molecular screening
- OI patients
  Interventions: Diagnostic Test: NGS molecular screening

INTERVENTIONS:
Diagnostic Test: NGS molecular screening

SUMMARY:
The coming out of Next Generation Sequencing (NGS) technologies, with documented advantages and reduced costs respect to Sanger sequencing, has provided new appealing approaches to diagnostic testing. Despite this, its use for routine diagnostic purposes requires certification in terms of reliability, as well as a cost-effectiveness evaluation.

To test the feasibility of using the Ion Torrent Personal Genome Machine (PGM) in clinical diagnosis, we assessed its performance to detect point mutations and big rearrangements previously identified with standard techniques. The diagnostic accuracy and the cost-effectiveness will be evaluated by Health Technology Assessment (HTA) analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Osteochondroma
* Clinical diagnosis of Osteogenesis Imperfecta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 400 DNA samples coming from MO and OI patients (including either dominant and recessive forms) will be included in the study (250 affected by MO and 150 by OI).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the accuracy of the Ion Torrent PGM platform for genetic variant detection (Diagnostic sensitivity evaluation) | at 30 months
  The accuracy of the Ion Torrent Personal Genome (PGM) to identify disease-causing mutations in patients affected by Multiple Osteochondromas (MO) and Osteogenesis Imperfecta (OI) needs to be validated for its routine diagnostic clinical use. To asses this, we will compare results obtained with the new NGS approach with those previously obtained with standard techniques (DHPLC/Sanger + MLPA) in a number of MO and OI patients.
HTA analysis to assess the cost-effectiveness, organizational and social implications of a screening strategy based on the IonPGM platform | at 36 months
  To demonstrate the pertinence in the use of this innovative technology in health care, we will examine the medical, social and economic implications according with Health Technology Assessment (HTA), a multi-disciplinary field of policy analysis applied to many different health care technologies before their diffusion and use. HTA aims at evaluating the real effectiveness of medical interventions, their proper use, access criteria and qualitative improvements, the clinical and organizational benefits, therefore suggesting how to manage, promote and discourage them.

IPD SHARING:
Plan to Share IPD: No
No plan